CLINICAL TRIAL: NCT00000218
Title: Pharmacotherapy and Intensive Treatment
Brief Title: Pharmacotherapy and Intensive Treatment - 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: NIDA-06954-2; R18-06954-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Carbamazepine

INTERVENTIONS:
Drug: Carbamazepine

SUMMARY:
The purpose of this study is to evaluate desipramine and carbamazepine in reducing cocaine craving; increase outpatient treatment capacity and evaluate their incidence of psychiatric disorders.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 353
Dates: Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Severity addiction
Depression
Depression, anxiety

CONTACTS AND LOCATIONS:
Overall Officials: William Haning, M.D., Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Kansas City, Missouri, United States